CLINICAL TRIAL: NCT00306800
Title: A Multicenter, Double Blind, Vehicle-Controlled, Randomized Study of Photodynamic Therapy (PDT) With Metvix 160 Mg/g Cream and Aktilite CL128 LED Light in Patients With Multiple Actinic Keratosis on the Face and/or Scalp
Brief Title: Metvix PDT Versus Vehicle PDT With Aktilite CL128 Lamp in Patients With Actinic Keratosis on the Face and Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC T404/05
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2010-09

CONDITIONS: Actinic Keratosis
Keywords: Methyl aminolevulinate; Photodynamic therapy; Aktilite CL128 LED light source; Multiple Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy

INTERVENTIONS:
Procedure: Photodynamic therapy with methyl aminolevulinate cream

SUMMARY:
The purpose of this study is to compare the efficacy of Photodynamic Therapy (PDT) with methyl aminolevulinate (MAL) cream to PDT with vehicle cream, using the the LED light source Aktilite CL128, in treatment of patients with multiple actinic keratosis (sun-damaged skin) on the face and / or scalp

DETAILED DESCRIPTION:
Actinic keratoses are pre-malignant skin lesions, which may develop to squamous cell carcinomas (SCC). They are usually small, thin, erythematous, de-squamating lesions on light exposed atrophic skin and the lesions are often multiple.

Photodynamic therapy (PDT) is the selective destruction of abnormal cells through light activation of a photosensitiser in the presence of oxygen. These cells accumulate more photosensitiser than normal cells. The photosensitiser generates reactive oxygen species upon illumination.

For skin diseases, such as actinic keratosis (AK), there has been an increasing interest in using topically applied precursors of the photoactive porphyrins (PAP). The most commonly used precursors have been 5-aminolevulinic acid (ALA) and its derivatives. The present test drug contains methyl aminolevulinate, which penetrates the lesions well and shows high lesion selectivity.

Different light sources (i.e. CureLight, Aktilite CL16 and Aktilite CL128) have been used for the activation of PAP, which absorbs light in the range of 400-700 nm. The present study uses the Aktilite CL 128 lamp. Aktilite 128 is based on LED technology and emits a narrow red light spectrum with an average wavelength of 630 (+/-5) nm. This study is similar to two other studies performed, on which the U.S. approval of Metvixia® cream is based except for the light source used. This study is one of two studies performed to document the safety and efficacy of the Aktilite CL 128 lamp when used in combination with Metvixia® cream.

Previous studies have shown that the risks attributed to Metvixia® PDT are few and related mainly to transient pain and local erythema during and shortly after treatment. These reactions are part of the expected local phototoxicity reaction. PDT offers an advantage to other treatment modalities for actinic keratosis, being a non-invasive treatment available on an outpatient basis. Several separate lesions can be treated simultaneously and the same lesion(s) can be treated repeatedly with success. There are no known systemic toxicity or interaction with other medication. The treatment is also lesion selective, leaving the surrounding tissue intact and functional, also allowing excellent cosmetic results after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of 4-10 previously untreated, not pigmented, non-hyperkeratotic AK lesions of 3 mm or more diameter of Grade 1 and/or 2 of the face and/or scalp where other therapies are unacceptable or considered medically less appropriate.
* Males or females above 18 years of age.
* Written informed consent

Exclusion Criteria:

* Patients with porphyria.
* Patients immunosuppressed for idiopathic, disease specific or therapeutic reasons.
* Known allergy to MAL, a similar PDT compound or excipients of the cream.
* Patients with history of hypersensitivity to nut products or other known protein antigens.
* Participation in other clinical studies either currently or within the last 30 days.
* Patients receiving local treatment (including cryotherapy and curretage) in face / scalp area within the last 30 days.
* Patients receiving topical treatment (including imiquimod, 5-FU and diclofenac) in face / scalp area within the last 3 months.
* Pregnant or breast-feeding: All women of child-bearing potential must use adequate contraception (oral contraceptives, intrauterine device, contraceptive skin patch, etc) during the treatment period and one month thereafter. In addition, they must have a negative pregnancy test prior to treatment.
* Any conditions that may be associated with a risk of poor protocol compliance.
* Patients currently receiving regular ultraviolet radiation therap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-09; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Primary: Primary outcome: To compare the patient complete response rate of MAL PDT to that of vehicle PDT 3 months after the last treatment in patients with multiple actinic keratoses on the face and/or scalp

SECONDARY OUTCOMES:
Secondary: The secondary outcomes: To compare local Adverse Events (treatment site Adverse Events (AEs) between MAL PDT and vehicle PDT; To compare the lesion complete response rate between MAL PDT and vehicle PDT 3 months after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Pariser, MD, Principal Investigator — Virginia Clinical Research
Locations (7):
- United States (7):
  - Spencer Dermatology and Skin Surgery, St. Petersburg, Florida
  - Laser and Skin Surgery Center, New York, New York
  - Dermatology Associates of Rochester, Rochester, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Dermresearch Inc, Austin, Texas
  - Texas Dermatology Research Institute, Dallas, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas

REFERENCES:
- [Background] Pariser DM, Lowe NJ, Stewart DM, Jarratt MT, Lucky AW, Pariser RJ, Yamauchi PS. Photodynamic therapy with topical methyl aminolevulinate for actinic keratosis: results of a prospective randomized multicenter trial. J Am Acad Dermatol. 2003 Feb;48(2):227-32. doi: 10.1067/mjd.2003.49. PMID 12582393
- [Background] Freeman M, Vinciullo C, Francis D, Spelman L, Nguyen R, Fergin P, Thai KE, Murrell D, Weightman W, Anderson C, Reid C, Watson A, Foley P. A comparison of photodynamic therapy using topical methyl aminolevulinate (Metvix) with single cycle cryotherapy in patients with actinic keratosis: a prospective, randomized study. J Dermatolog Treat. 2003 Jun;14(2):99-106. doi: 10.1080/09546630310012118. PMID 12775317